CLINICAL TRIAL: NCT01670214
Title: A Randomized, Placebo-control of Pulsed Electromagnetic Field Therapy as Preventive Treatment of Refractory Migraine
Brief Title: Pulsed Electromagnetic Field Therapy in the Refractory Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Niyayesh Clinic (Other)
Collaborators: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Boshra Hatef, Phd student of physiotherapy, Tarbiat Modarres University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIYAYESH CLINIC 1
Record Dates: First submitted 2012-01-24; First posted 2012-08-22 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2012-08

CONDITIONS: Refractory Migraine
Keywords: RM; R-CM; based on ICHD-2 criteria
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pulsed electromagnetic field (Active Comparator): parameters of the pulsed electromagnetic field are frequency:10 Hz, intensity 4-5 mT, 6 sessions phase 1 treatment and added 6 sessions for phase 2 treatment (3 sessions per week)
  Interventions: Procedure: pulsed electromagnetic field
- pulsed electromagnetic field (Placebo Comparator): patients are placed under off instrument while who is kept blind to know it for 6 sessions (3 sessions per week).
  Interventions: Procedure: pulsed electromagnetic field

INTERVENTIONS:
Procedure: pulsed electromagnetic field — parameters of the pulsed electromagnetic field are frequency:10 Hz, intensity 4-5 mT, 6 sessions( 2 week) for placebo and phase 1 treatment ( 3 sessions in week) and added 6 sessions for phase 2 treatment. the solenoid diameter of instrument is 70 cm is placed around the head.

SUMMARY:
Pulsed electromagnetic field (PEMF) as prophylactic treatment may prevent the attacks of migraine or decrease them even in the patients with refractory migraine.

DETAILED DESCRIPTION:
Migraine is most common among patients who seek medical care for headache. The prevalence of migraine is around 10 % in Iran. The many studies of migraine pathophysiology imply that the brain of migraine patient is impaired in term of cerebral circulation and baseline activity of brain stem, monoaminergic system and cortex. Then headache is only a sign of the changes that occur in the brain to rid hazardous conditions. Based on this theory many electrophysiological and imaging abnormalities that were appeared in the brain before the aura or the headache were diminished in the early phases of the attack. It means the changes concurrent with headache are associated with a quasi normalization of cortical information processing. The different pharmacological and non-pharmacological treatments have proposed for migraine management. But some patients do not satisfactorily respond to or cannot tolerate current evidence-based treatments. This group of patients is often said to have refractory migraine (RM). Thus according to the enigmatic pathophysiology of migraine, a comprehensive treatment that affected all contributing factors in the migraine with minimal side effects is not provided yet.

Extremely low frequency magnetic fields (ELF MFs) as non-pharmacological treatment of migraine had good effect with weak evidence in the control of migraine. Recently based on extensive studies in the bioeffects of the low frequency electromagnetic field we can hope that this method can respond to many human disorders is unsolvable. The purpose of this study is to apply the best effective treatment protocol of ELF-MF on brain and circulatory system is extracted by using the latest findings of studies of low-frequency electromagnetic fields as intervention and apply it for refractory migraine patients in the form of a randomized one-blind placebo- controlled trial study. The evaluation of interventions is done subjectively (migraine dairy and MIDAS). Also we consider follow up period to confirm results.

ELIGIBILITY:
Inclusion Criteria:

Primary Diagnosis A. ICHD-II migraine or chronic migraine Refractory B. Headaches cause significant interference with function or quality of life despite modification of triggers, lifestyle factors, and adequate trials of acute and preventive medicines with established efficacy.

1. Failed adequate trails of preventive medicines, alone or in combination from at least 2 of 4 drug classes:

   * Beta-blockers
   * Anticonvulsants
   * Tricyclics
   * Calcium channel blockers
2. Failed adequate trials of abortive medicines from the following classes, unless contraindicated:

   * Both a triptan and DHE intranasal or injectable formulation
   * Either nonsteroidal anti-inflammatory drugs or combination analgesics
   * Adequate trial Period of time during which an appropriate dose of medicine is administered, typically at least 2 months at optimal or maximum-tolerated doses, unless terminated early due to adverse effects
   * Modifiers With or without medication overuse, as defined by ICHD-2
   * With significant disability, as defined by MIDAS > 11
   * [DHE = dihydroergotamine; ICHD = International Classification of Headache Disorders;MIDAS = Migraine Disability Assessment]
   * The prophylactic medications have been discontinued at least one month prior to enrollment

Exclusion Criteria:

* pregnancy
* epilepsy
* malignancy

Ages: 17 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
MIDAS | 6 months
  migraine disability score
headache frequency | 4 months
headache duration | 4 months
headache intensity | 4 months

SECONDARY OUTCOMES:
medications | 4 months
missed work | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Boshra Hatef, Phd student PT,TMU, Principal Investigator — Niyayesh Clinic; mansoore toghae, prof. neurology,TUMS, Study Director — sina hospital of Medical Science University of Tehran
Locations (1):
- Niyayesh clinic, Tehran, Iran

REFERENCES:
- [Background] B Hatef, B Majdoleslam, M Toghae, F Hashemirad. The Prophylactic Treatment of PEMF in the Refractory Migraine Headache, Double-Blind, Parallel Placebo-Controlled Study. CEPHALALGIA 33(s8): 98-99, 2013
- [Result] Boshra Hatef, Fahime Hashemirad, Gholam Hossein Meftahi, Leila Simorgh, Soodeh Razeghi Jahromi, Forough Rahimi, Mansoureh ToghaThe efficiency of pulsed electromagnetic field in refractory migraine headaches: a randomized, single-blinded, placebo-controlled, parallel group. international journal of clinical trial 3(1): 24-31, 2016
- See also: Related Info — http://www.ijclinicaltrials.com/index.php/ijct/article/view/99